CLINICAL TRIAL: NCT06024850
Title: Predictive Factors of Good Results After Multiligamentar Knee Reconstruction (MLKR)
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN342022/CHUSTE
Record Dates: First submitted 2023-07-21; First posted 2023-09-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Knee Ligament Injury
Keywords: Multiligamentar; injury; knee; magnetic resonance imaging (MRI); knee reconstruction; knee dislocation
MeSH Terms: conditions — Wounds and Injuries; Knee Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiligamentar knee reconstruction: Any patient who benefits of a multiligamentar knee reconstruction at hospital of Saint-Etienne will be included.
  Datas collected by medical record.
  Interventions: Other: Datas collected

INTERVENTIONS:
Other: Datas collected — Datas collected by medical record: medical data (weight, height, smoking status, history) and socio-demographic data (age, occupation, type of injury) information, assessment of knee function before surgery, at 6 months and 1 year after surgery, magnetic resonance imaging (MRI) and radiological imaging at 1 year after surgery, results of the Iso-kinetic Muscle Assessment Test at 1 year after surgery to objectively determine the recovery of muscle function
  The data collected will be used to perform a statistical analysis to evaluate the factors predicting a good long-term post-surgical evolution

SUMMARY:
Multiligamentar knee injury has consequences on knee function (instability, arthritis, life disagreement). Surgical reconstructions have known recent evolutions. The goal of this study is to evaluate functional and clinical results at one year of those new surgical technics. A clinical and functional follow up will be performed before the surgery, then at 6 months and one year.

DETAILED DESCRIPTION:
Patients will also benefit of a Magnetic Resonance Imaging (MRI) and isokinetic evaluations at one year.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who benefits of a multiligamentar knee reconstruction at hospital of Saint-Etienne

Exclusion Criteria:

* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who benefits of a multiligamentar knee reconstruction at hospital of Saint-Etienne will be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Functional score : International Knee Documentation Committee (IKDC) | Months : 0, 6 and 12
  The International Knee Documentation Committee (IKDC) is a questionnaire that assigns patients an overall functional score. Three categories are examined by the questionnaire: symptoms, sports activity and knee function, on a scale of 0 to 100.

SECONDARY OUTCOMES:
Functional score : Knee Injury and Osteoarthritis Outcome Score (KOOS) | Months : 0, 6 and 12
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is used to assess immediate and long-term patient outcomes after knee injury. Five outcomes are assessed by the self-administered KOOS: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life, on a scale of 0 to 100.
Visual Analogue Scale (VAS) scale | Months: 0, 6 and 12
  Analysis of the Visual Analogue Scale (VAS) scale (from 0 to 10, 10 = pain ++)
Laxity | Month : 12
  Laxity assessed by Magnetic Resonance Imaging (MRI)
Joint amplitudes | Months: 0, 6 and 12
  Joint amplitudes assessed by the iso-cinetic test
Clinical data | Month : 0
  Data collected at inclusion
Recovery of muscle function | Month : 12
  Recovery of muscle function measured by iso kinetic muscle assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas NERI, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No